CLINICAL TRIAL: NCT02927587
Title: Optimal TCI Regimen for Sedation of Elderly Undergoing Fiberoptic Bronchoscopy: A Prospective Randomized Controlled Trial.
Brief Title: Optimal TCI Regimen for Sedation of Elderly Undergoing Fiberoptic Bronchoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: brofiber
Record Dates: First submitted 2016-10-03; First posted 2016-10-07 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Adverse Effects
Keywords: TCI; fiberoptic bronchoscopy; sedation
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- The induction Cet of propofol 1 (Experimental): The induction Cet of propofol was targeted at 1 ug/ml.
  Interventions: Drug: The induction Cet of propofol
- The induction Cet of propofol 2 (Other): The induction Cet of propofol was targeted at 2 ug/ml.
  Interventions: Drug: The induction Cet of propofol

INTERVENTIONS:
Drug: The induction Cet of propofol — The induction Cet of propofol was targeted respectively at 1 and 2 ug/ml.
  Other Names: propofol

SUMMARY:
Target-Controlled Infusion (TCI) of Propofol has been proved to be a safe agent for conscious sedation in flexible bronchoscopy (FB) .However, the target setting of "effect-site" concentration (Cet) of propofol is still unclear in the elderly population .The aim of this study was to compare two induction Cet of propofol in elderly patients undergoing flexible bronchoscopy.

DETAILED DESCRIPTION:
BACKGROUND:Bronchoscopy is nowadays a very common and widespread technique that allows the physician to proceed for both diagnostic and therapeutic interventions. The risks of this procedure are low and depend mostly on the health of the patient. In our study we only considered the elderly ( age > 65 years old) which makes the risks even higher.

Target-Controlled Infusion (TCI) of Propofol has been proved to be a safe agent for conscious sedation in flexible bronchoscopy (FB) due to its fast onset of action and rapid recovery time. By virtue of an aging population, the number of bronchoscopy performed will likely increase in the elderly patients , however, the target setting of "effect-site"concentration (Cet) of propofol is still unclear among this population.

The aim of this study was to compare two induction Cet of propofol in elderly patients undergoing flexible bronchoscopy.

METHODS: Seventy patients were randomly divided into 2 groups . All patients were of American Society of Anesthesiologists (ASA) physical status of I-III, aged more than 65 years old and between 45 and 100 kg in weight. The induction Cet was targeted respectively at 1 and 2 ug/ml. Upon reaching the modified observer's assessment of alertness/sedation(MOAA/S) score 0-3, the Cet was increased or reduced during the procedures and the Ce level was set for the maintenance of sedation. Induction time, diagnostic procedures as well as the occurrence of adverse events such as apnea , hypotension or hypertension, heart rate, oxygen saturation (SpO2) ,any cardiac event, cough score, frequency of adjustments of drug doses were recorded.

The patient will be monitored during the procedure with periodic blood pressure checks, respiratory rate, continuous electrocardiogram monitoring of heart and oxygen measurement.

ELIGIBILITY:
Inclusion Criteria:

* body mass index < 30 in males or <28 in females
* an ASA physical status I and III

Exclusion Criteria:

* severe sleep apnoea syndrome (apnoea-hypopnea index > 40)
* bradycardia
* hypotension

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-11; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
the adverse events(apnea , hypotension or hypertension, heart rate, oxygen saturation ,any cardiac event, cough score) | 1 and 2 hours
  Change from beginning of sedation to removal of bronchoscope

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Dalian Medical University, Dalian, Liaoning, China